CLINICAL TRIAL: NCT01689090
Title: Diameter Changes of Retinal Vessels During Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HypNOCOX
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2015-08

CONDITIONS: Diabetes Mellitus Type 1; Diabetic Maculopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Cyclooxygenase Inhibitors; omega-N-Methylarginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoxia (Experimental): Inhaling hypoxic gas mixture to induce hypoxemia during recordings of diameter changes of retinal vessels. Recording are performed during hypoxia alone and in combination with the associated interventions at two examination days.
  Interventions: Other: COX inhibitor; Other: L-NG-monomethyl arginine citrate; Other: COX inhibitor + L-NG-monomethyl arginine citrate
- Normoxia (Experimental): Breathing atmospheric air during recordings of diameter changes of retinal vessels. Recording are performed during normoxia alone and in combination with the associated interventions at two examination days.
  Interventions: Other: COX inhibitor; Other: L-NG-monomethyl arginine citrate; Other: COX inhibitor + L-NG-monomethyl arginine citrate

INTERVENTIONS:
Other: COX inhibitor — Administration of 1 drop voltaren 45 minutes before recordings of diameter changes of retinal vessels are initiated
  Other Names: Eye drops voltaren 1 mg/ml
Other: L-NG-monomethyl arginine citrate — Intravenous administration of L-NMMA during recordings of diameter changes of retinal vessels
  Other Names: L-NMMA
Other: COX inhibitor + L-NG-monomethyl arginine citrate — Combination of interventions. Administration of an eye drop voltaren and 45 minutes later infusion with L-NMMA is started and recording of diameter changes of retinal vessels is performed

SUMMARY:
The primary objective is to study if an inhibition of nitric oxide and/or prostaglandins affect the diameter changes of retinal vessels observed during hypoxia. Diameter changes are studied using the Dynamic Vessel Analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 1 without retinopathy
* Diabetic retinopathy

Exclusion Criteria:

* Cardio-vascular disease
* Lung disease
* Pregnancy
* Previous ocular disease other than retinal branch vein occlusion
* Previous treatment with medications influencing on the intraocular pressure or the metabolism of nitric oxide or prostaglandins

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Diameter changes of retinal vessels | Examination day 1 and 2
  Comparing the differences of diameter changes occuring during each of the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Line Pedersen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Ophthalmology, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Petersen L, Bek T. Post-hypoxic constriction of retinal arterioles is impaired during nitric oxide and cyclo-oxygenase inhibition and in diabetic patients without retinopathy. Graefes Arch Clin Exp Ophthalmol. 2017 Oct;255(10):1965-1971. doi: 10.1007/s00417-017-3746-2. Epub 2017 Jul 27. PMID 28752370
- [Derived] Petersen L, Bek T. The diameter response of retinal arterioles in diabetic maculopathy is reduced during hypoxia and is unaffected by the inhibition of cyclo-oxygenase and nitric oxide synthesis. Graefes Arch Clin Exp Ophthalmol. 2016 Dec;254(12):2339-2346. doi: 10.1007/s00417-016-3399-6. Epub 2016 Jun 7. PMID 27270566